CLINICAL TRIAL: NCT03687047
Title: Evaluation the Impact of the Use of New Complete Denture (Prothesis) on the OHRQoL in Total Edentulous Patients Comparing to Dentate Individuals
Brief Title: Impact of the Use of New Complete Denture on the Oral Health Related to Quality of Life (OHRQoL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Livia Azeredo Alves Antunes, Clinical professor, Universidade Federal Fluminense
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Complete denture and OHRQoL
Record Dates: First submitted 2018-09-20; First posted 2018-09-27 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Edentulous Jaw; Quality of Life
Keywords: DENTADURES; EDENTULOUS; MASTIGATORY PERFORMANCE
MeSH Terms: conditions — Jaw, Edentulous; Mouth, Edentulous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New complete dentures (Experimental): Steps: 1) Preliminary impressions will be done using stock trays and impression compound; 2) primary casts will be fabricated to make custom trays for definitive impressions; 3) definitive impressions will be made using zinc oxide eugenol impression paste;4) definitive impressions will be poured with type III dental stone to obtain mastercasts; 5)jaw relations will be recorded, and the casts will be mounted on the articulator; 6) the artificial acrylic resin teeth will be arranged, esthetics will be verified, and the trial dentures will be flasked and polymerized (72°C per 12 hours). The dentures will be finished and polished for insertion and follow-up. After denture insertion, post-denture insertion instructions such as oral hygiene will be explained to the patients.
  The Oral Health Related to Quality of Life assessment will be conducted before treatment (Baseline) and at 3, 6, 9, 12 months after treatment.
  Interventions: Device: New complete dentures

INTERVENTIONS:
Device: New complete dentures — Preliminary impressions using stock trays and impression compound; primary casts fabricated to make custom trays for definitive impressions; definitive impressions using zinc oxide eugenol impression paste; definitive impressions poured with type III dental stone to obtain mastercasts; jaw relations will be recorded, and the casts will be mounted on the articulator; the artificial acrylic resin teeth will be arranged, esthetics will be verified, and the trial dentures will be flasked and polymerized (72°C per 12 hours). The dentures will be finished and polished for insertion and follow-up.

SUMMARY:
The aim of this project was to evaluate the impact before and after (3, 6, 9, and 12 months) of oral rehabilitation with conventionalof the insertion of new complete dentures (CD) in the oral health-related quality of life (OHRQoL) in total edentulous patients compared to dentate individuals. This is a clinical trial study approved by the Research Ethics Committee (nº 31105714.7.0000.5626 ) which was conducted on 122 patients who attended the clinics of Federal Fluminense University, with the necessity of CD. The eligibility criteria were: healthy patients without disabilities; aged up to 50 years; complete upper and or lower jaw edentulism for a minimum 5 years; the presence of adequate healthy tissue to support the prosthesis; adequate cognitive ability and understanding to respond to the questions posed. It will be excluded patient with motor disabilities, cognitive impairment and people with special needs. After the installation of the CD a follow-up of one week, three, six, nine, twelve and eighteen months will be performed. The Oral Health Impact Profile (OHIP-Edent) instrument will be applied (in form of an interview) to evaluate the impact of CD on OHRQoL. The scores of the OHIP-Edent index will be calculated using the additive method, summing the numeric response codes for each item. Shapiro-Wilk test revealed nonparametric distribution of data. Chi-square, Mann-Whitney U, and Kruskal-Wallis tests were performed for comparing groups according to sociodemographic data. Kruskal-Wallis test was per- formed for comparing groups and treatments throughout time. A significance level of 5% was adopted, and all analyses were performed on Statistical Analysis System (SAS) version 9.3 software. The responsiveness was assessed by analyzing the change of the scores on the scales and subscales. The changes was calculated by subtracting the post-treatment scores from the before-treatment scores. Positive change scores will indicate an improvement in OHRQoL, while negative scores will indicate deterioration.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients without disabilities;
* aged up to 50 years;
* patient with complete upper and or lower jaw edentulism for a minimum 5 years;
* patient with presence of adequate healthy tissue to support the prosthesis;
* patient with adequate cognitive ability and understanding to respond to the questions posed

Exclusion Criteria:

* patient with motor disabilities;
* patient with cognitive impairment
* people with special needs.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of oral heath related to quality of life from edentulous patient after use new complete denture | 12 MESES
  After the installation of the new prothesis (complete denture) a follow-up (one week, three, six, nine, twelve months) will be performed. The Oral Health Impact Profile (OHIP-Edent) instrument will be applied (in form of interview) to evaluate the impact of new prothesis (complete denture) on OHRQoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal Fluminense, Nova Friburgo, Rio de Janeiro, Brazil